CLINICAL TRIAL: NCT00661076
Title: A Randomized, Open Label Study to Compare the Effect of Combination Treatment With PEGASYS + Adefovir Dipivoxil Versus PEGASYS Monotherapy on HBV-DNA and ALT Levels in Patients With HBeAg-negative, Chronic Hepatitis B.'
Brief Title: ADVANCE Study: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) + Adefovir Dipivoxil in Patients With Hbe(-) Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20622
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; peginterferon alfa-2a

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: adefovir dipivoxil; Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: adefovir dipivoxil; Drug: peginterferon alfa-2a [Pegasys]
- 3 (Active Comparator)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: adefovir dipivoxil — 10mg po daily for 96 weeks (arm 1) or 48 weeks (arm 2)
  Arms: 1; 2
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms weekly for 48 weeks

SUMMARY:
This 3 arm study will compare the efficacy and safety of combination therapy with PEGASYS + adefovir dipivoxil (ADV) versus PEGASYS monotherapy, in HBeAg-negative chronic hepatitis B patients.Patients will be randomized to receive 1)PEGASYS 180 micrograms sc weekly + ADV 10mg po daily for 48 weeks, followed by ADV 10mg po monotherapy for an additional 48 weeks, and a further 48 week treatment-free follow-up, 2)PEGASYS 180 micrograms sc weekly + ADV 10mg po daily for 48 weeks, followed by a 96 week treatment-free follow-up, or 3)PEGASYS 180 micrograms sc monotherapy weekly for 48 weeks, followed by a 96 week treatment-free follow-up. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* chronic hepatitis B;
* positive HBsAg, positive anti-HBe, negative anti HBsAg, negative HBeAg for at least the prior 6 months;
* either nucleoside analogue naive, or has not received IFN-a in the past 6 months.

Exclusion Criteria:

* positive for hepatitis A, C, D or HIV;
* history or other evidence of a medical condition associated with chronic liver disease other than hepatitis B;
* antiviral, antineoplastic or immunomodulatory treatment <=6 months prior to first dose of randomized treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Normalization of ALT, and HBV-DNA <400 copies/mL | Week 96 for arm 1; week 48 for arms 2 and 3
HBsAg quantitative loss and anti-HBs seroconversion | Weeks 48, 96 and 144

SECONDARY OUTCOMES:
AEs, lab parameters, vital signs | Throughtout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara
  - Gaziantep